CLINICAL TRIAL: NCT07051655
Title: The Effects of Exogenous Ketones on Cognitive Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Katherine Sweatt, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300013940; UAB (Other: UAB)
Record Dates: First submitted 2025-06-03; First posted 2025-07-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Placebo - Control; Ketone Monoester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will undergo two test days (Test Day 1 and Test Day 2) separated by 3-7 days. On one test day, participants will consume a single dose of placebo (357 mg/kg of body weight). Thirty minutes after consuming the placebo, cognitive assessments will be completed including NIH Toolbox cognitive assessments, Senaptec Sensory Station, and driving simulation.
  Interventions: Dietary Supplement: Placebo
- ketone monoester (KME) (Experimental): Participants will undergo two test days separated by 3-7 days. On one test day, participants will consume a single dose of ketone monoester (KME) (357 mg/kg of body weight). Thirty minutes after consuming the KME, cognitive assessments will be completed including NIH Toolbox cognitive assessments, Senaptec Sensory Station, and driving simulation.
  Interventions: Dietary Supplement: Ketone Monoester (KE)

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE) — Participants will undergo two test days separated by 3-7 days. On both test days, participants will arrive fasted and consume a single dose of ketone monoester or placebo (357 mg/kg of body weight) in random order. Drinks will be prepared by non-study personnel and matched in taste, texture, and appearance to maintain blinding. Thirty minutes after consuming the ketone monoester or placebo, cognitive assessments will be completed including NIH Toolbox cognitive assessments, Senaptec Sensory Station, and driving simulation.
  Other Names: ketone monoester (KME)
  Arms: ketone monoester (KME)
Dietary Supplement: Placebo — Participants will undergo two test days separated by 3-7 days. On one test day, participants will consume a single dose of placebo (357 mg/kg of body weight). Thirty minutes after consuming the placebo, cognitive assessments will be completed including NIH Toolbox cognitive assessments, Senaptec Sensory Station, and driving simulation.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the acute effects of exogenous ketone monoester (KME) supplementation on cognitive function in three groups of adults aged 19-55 years: (1) obese, sedentary individuals; (2) lean, sedentary individuals; and (3) lean individuals who engage in regular physical activity (e.g., collegiate or amateur athletes). The main questions it aims to answer are to:

* Assess the effects of acute KME supplementation versus placebo on cognitive, sensorimotor, and functional outcomes within groups.
* Compare cognitive performance across the three groups.

The primary outcome is cognitive performance assessed using the NIH Toolbox Cognition Battery. Secondary Outcomes include sensorimotor performance, measured using the Senaptec Sensory System, and driving performance, assessed with a driving simulator.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the acute effects of exogenous ketone monoester (KME) supplementation on cognitive function in three groups of adults aged 19-55 years: (1) obese, sedentary individuals; (2) lean, sedentary individuals; and (3) lean individuals who engage in regular physical activity (e.g., collegiate or amateur athletes).

Exogenous ketones are considered a functional food, providing potential health benefits beyond basic nutrition. Specifically, KME has been shown to elevate circulating β-hydroxybutyrate (βHB), an alternative brain fuel that may enhance cognitive performance. Prior studies have demonstrated that KME improves cognition in individuals with Alzheimer's disease and mild cognitive impairment; however, its effects in otherwise healthy, sedentary individuals-particularly those with obesity-or in physically active individuals remain unknown.

Emerging evidence suggests that individuals with obesity may exhibit early cognitive deficits, especially in executive function and processing speed, which could increase their risk of accelerated cognitive decline with aging. These deficits may be partially attributed to impaired cerebral glucose metabolism. Since ketones serve as an efficient alternative energy substrate for the brain, ketone supplementation may help compensate for these metabolic deficits and enhance cognitive performance.

This study aims to compare cognitive performance across the three groups and assess the effects of acute KME supplementation versus placebo on cognitive, sensorimotor, and functional outcomes. The primary outcome is cognitive performance assessed using the NIH Toolbox Cognition Battery. Secondary Outcomes include sensorimotor performance, measured using the Senaptec Sensory System, and driving performance, assessed with a driving simulator.

This three-group design allows for the investigation of differential responses to ketone supplementation across a spectrum of metabolic health and physical conditioning. By using sensitive, multimodal assessment tools, this study will help determine whether exogenous ketones confer cognitive and functional benefits broadly, or whether these effects are most pronounced in metabolically impaired populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-55 years
* BMI 30-40 (obese group) or 18-25 (lean and athlete groups)
* Sedentary status (<2 hrs/week of structured physical activity) for obese and lean groups
* Active athlete status (≥5 days/week of structured activity) for athlete group

Exclusion Criteria:

* Diagnosed neurological conditions (e.g., Parkinson's disease, multiple sclerosis, schizophrenia, muscular dystrophy, stroke, cerebral palsy)
* History of seizures
* Use of medications for diabetes, mood disorders, or attention disorders
* Pregnant or breastfeeding
* Current or recent use (within 1 month) of exogenous ketone supplements or adherence to a ketogenic diet

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox Cognition Battery Composite Score and Domain-Specific Subtests - Executive function | Test Day 1 and Test Day 2
  Cognitive function will be assessed using the NIH Toolbox Cognition Battery, administered on an iPad.
  - Dimensional Change Card Sort Test - Measures executive function and cognitive flexibility by assessing the ability to switch between mental rules.
NIH Toolbox Cognition Battery Composite Score and Domain-Specific Subtests - Attention | Test Day 1 and Test Day 2
  Cognitive function will be assessed using the NIH Toolbox Cognition Battery, administered on an iPad.
  - Flanker Inhibitory Control and Attention Test - Evaluates attention and the ability to inhibit responses to distracting information.
NIH Toolbox Cognition Battery Composite Score and Domain-Specific Subtests - Processing Speed | Test Day 1 and Test Day 2
  Cognitive function will be assessed using the NIH Toolbox Cognition Battery, administered on an iPad.
  - Oral Symbol Digit Substitution Test - Assesses processing speed by requiring participants to match symbols and digits under time pressure.
NIH Toolbox Cognition Battery Composite Score and Domain-Specific Subtests - Memory | Test Day 1 and Test Day 2
  Cognitive function will be assessed using the NIH Toolbox Cognition Battery, administered on an iPad.
  - Picture Sequence Memory Test - Tests episodic memory by having participants recall sequences of illustrated scenes in the correct order.

SECONDARY OUTCOMES:
Senaptec Sensory Station - Visual Acuity | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station. This includes:
  Visual Clarity Test - Measures the sharpness of vision using high-contrast letters; similar to a Snellen chart.
Senaptec Sensory Station - Visual perception | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Contrast Sensitivity - Assesses ability to detect subtle differences in luminance; important in low-light or low-contrast environments.
Senaptec Sensory Station - Stereopsis, spatial awareness | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Depth Perception - Measures the ability to judge the relative distance between objects using binocular vision.
Senaptec Sensory Station - Oculomotor control | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Near-Far Quickness - Assesses speed and accuracy in shifting focus between near and far objects; linked to accommodative and vergence flexibility.
Senaptec Sensory Station - Visual search | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Target Capture - tests speed and accuracy in identifying and responding to a target among distractors.
Senaptec Sensory Station - Visual working memory | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Perception Span - Evaluates ability to recall the location and identity of briefly presented visual stimuli.
Senaptec Sensory Station - Attention | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Go/No-Go - Assesses impulse control by requiring responses to specific stimuli while inhibiting others
Senaptec Sensory Station - Processing Speed | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Reaction Time - Measures the speed of motor response to a visual stimulus; includes both simple and choice RT.
Senaptec Sensory Station - Visual Tracking | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Multiple Object Tracking - Requires simultaneous tracking of multiple moving targets among distractors
Senaptec Sensory Station - Visuomotor Integration | Test Day 1 and Test Day 2
  Participants will complete the full suite of visual and sensorimotor evaluations within the "Evaluation" tab of the Senaptec Sensory Station.
  Eye-Hand Coordination - Measures the ability to synchronize visual input with precise hand movement.
Driving Simulator Performance Metrics - Attention | Test Day 1 and Test Day 2
  Cognitive and functional performance will be assessed using a high-fidelity driving simulator.
  - Lane-keeping variability
  Driving simulator data will provide an ecologically valid, real-world proxy of cognitive-motor integration and decision-making under time pressure.
Driving Simulator Performance Metrics - Reaction Time | Test Day 1 and Test Day 2
  Cognitive and functional performance will be assessed using a high-fidelity driving simulator. Participants will complete a standardized driving task
  * Mean reaction time to unexpected events (e.g., pedestrian crossing)
  * Braking accuracy and response latency
  Driving simulator data will provide an ecologically valid, real-world proxy of cognitive-motor integration and decision-making under time pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- 916 Building, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No